CLINICAL TRIAL: NCT00662389
Title: TP-1013 Pilot 1: Application of the Apsara Thermal Wand System
Brief Title: Application of the Apsara Thermal Wand System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Apsara Medical Corporation (Industry)
Responsible Party: Kim Tompkins, VP, Clinical/Regulatory/Quality
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEIRB08-090
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2009-08-28 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-07

CONDITIONS: Tightening of Skin Laxity
Keywords: skin laxity, wrinkles, rhytids
MeSH Terms: conditions — Cutis Laxa

ARMS (1):
- A (Experimental)
  Interventions: Device: Apsara Thermal Wand System

INTERVENTIONS:
Device: Apsara Thermal Wand System — Single radiofrequency cycle to dermal tissue

SUMMARY:
The purpose of this feasibility study is to gain an initial assessment of the acute safety and performance of the Apsara Thermal Wand System in human facial tissue.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoker
* Glogau class 1-3
* Previously chosen to undergo facelift

Exclusion Criteria:

* Pregnant, nursing
* Implanted electro-mechanical device
* Allergy to anesthesia or device metals
* Collagen vascular disease
* History of keloid or hypertrophic scar formation
* Uncontrolled diabetes
* Long term steroid or other immunologic inhibitor use
* Previous treatment to target area
* Does not consent to study
* Does not consent to photography or histological evaluation

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bryant A. Toth, MD, FACS, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A--Thermal Wand Application
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | A--Thermal Wand Application
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 61.7 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: Number of Serious Adverse Events
Time Frame: Immediate
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | A--Thermal Wand Application
Number analyzed (Participants) | 4
Number of Serious Adverse Events | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less